CLINICAL TRIAL: NCT02932956
Title: Glypican 3-specific Chimeric Antigen Receptor Expressed in Autologous T Cells as Immunotherapy for Patients With Pediatric Solid Tumors
Brief Title: Glypican 3-specific Chimeric Antigen Receptor Expressed in T Cells for Patients With Pediatric Solid Tumors (GAP)
Acronym: GAP
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); Cancer Prevention Research Institute of Texas (Other); The V Foundation (Other); Cookies for Kids' Cancer (Other); Curing Kids' Cancer Foundation (Other)
Responsible Party: Principal Investigator, David Steffin, MD, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-39410- GAP; GAP (Other: Baylor)
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Liver Cancer
Keywords: GPC3-CAR T cells; GPC3; Glypican; Liver cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Cyclophosphamide; fludarabine phosphate; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GAP T cells + Fludarabine and Cytoxan (Experimental): GPC3-Car (GAP T cells) along with lymphodepleting chemotherapy (Cytoxan and Fludarabine) will be administered to patients with GPC3-positive solid tumors.
  Interventions: Genetic: GAP T cells; Drug: Cytoxan; Drug: Fludara

INTERVENTIONS:
Genetic: GAP T cells — Five different dosing schedules will be evaluated. Three to six patients will be evaluated on each dosing schedule. The following dose levels will be evaluated:
  DL1: 1x10^7/m2
  DL2: 3x10^7/m2
  DL3: 1x10^8/m2
  DL4: 3x10^8/m2
  DL5: 1x10^9/m2
  The doses are calculated according to the actual number of GPC3-CAR transduced T cells.
  Other Names: GPC3-CAR T cells
Drug: Cytoxan — Cyclophosphamide will be given at a dose of 500 mg/m2/day for 3 days given intravenously.
  Other Names: Cyclophosphamide
Drug: Fludara — Fludarabine will be given at a dose of 30 mg/m2/day for 3 days given intravenously.
  Other Names: Fludarabine

SUMMARY:
This study enrolls patients who have GPC3-positive solid tumors currently. Patients may be considered if the cancer has come back, has not gone away after standard treatment or the patient cannot receive standard treatment. This research study uses special immune system cells called GAP T cells, a new experimental treatment.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells. Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat patients with cancers. They have shown promise, but have not been strong enough to cure most patients.

Investigators have found from previous research that they can put a new gene into T cells that will make them recognize cancer cells and kill them. In preclinical studies, the investigators made several genes called a chimeric antigen receptor (CAR), from an antibody called GC33 that recognizes glypican-3, a proteoglycan found on solid tumors including pediatric liver cancers (GPC3-CAR). This study will test T cells genetically engineered with a GPC3-CAR (GAP T cells) in patients with GPC3-positive solid tumors (currently only enrolling liver tumors).

The GAP T cells are an investigational product not approved by the Food and Drug Administration.

The purpose of this study is to find the biggest dose of GAP T cells that is safe, to see how long they last in the body, to learn what the side effects are and to see if the GAP T cells will help people with GPC3-positive solid tumors. This study enrolls patients who have GPC3-positive solid tumors (currently only enrolling liver tumors).

DETAILED DESCRIPTION:
Approximately 18-30 subjects will participate in the treatment part of this study.

Maximum of 180 mL of blood (not exceeding 3ml/kg/day) is collected from patients to grow the T cells and a retrovirus (a special virus that can insert the GPC3 CAR gene into the T cells) is used to genetically engineer them. After the CAR gene was put into the T cells, the investigators make sure that they are able to kill GPC3 positive solid tumor cells in the laboratory.

LYMPHODEPLETION CHEMOTHERAPY:

Several studies suggest that the infused T cells need room to be able to proliferate and accomplish their functions and that this may not happen if there are too many other T cells in circulation. Because of that, participants will receive treatment with cyclophosphamide (Cytoxan) and fludarabine for 3 days before receiving the T-cell infusion. These drugs will decrease the numbers of the participants' own T cells before the investigators infuse the GAP T CELLS.

WHAT THE INFUSION WILL BE LIKE:

After making these cells, they will be frozen. If the patient agrees to participate in this study, at the time the patient is scheduled to be treated, the cells will be thawed and injected into the patient over 5 to 10 minutes. The participant will receive the GAP T CELLS 48 to 72 hours after completing the chemotherapy.

This is a dose escalation study, which means that the investigators do not know the highest dose of GAP T cells that is safe. To find out, the investigators will give the cells to at least 3 participants at one dose level. If that is safe, the investigators will raise the dose given to the next group of participants. The dose each patient gets depends on how many participants get the agent before that patient and how they react. The investigator will tell each patient this information. This will help the participant think about possible harms and benefits. Since the treatment is experimental, what is likely to happen at any dose is not known.

All of the treatments will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital.

Medical tests before treatment:

* Physical exam and History
* Blood tests to measure blood cells, kidney and liver function.
* Pregnancy test (if the participant is a female who can get pregnant)
* If the participant is infected with the hepatitis B virus (HBV) the investigators will do a test to measure the levels of the virus
* Measurements of the participant's tumor by scans and the tumor marker alfa-fetoprotein (AFP), if the participant's tumor produces this protein.

Medical tests during and after treatment:

* Physical exams and History
* Blood tests to measure blood cells, kidney and liver function
* If the participant is infected with the hepatitis B virus (HBV) the investigators will repeat the test and monitor the levels of the virus
* Measurements of the participant's tumor by scans (4-6 weeks after the infusion) and AFP (if applicable at 1, 2, and 4 weeks after the infusion).
* Tumor biopsy between 2-4 weeks after the infusion and as clinically indicated thereafter. For additional clinically indicated tumor biopsies, investigators will ask for a portion of the sample for research.

FOLLOW-UP STUDIES

The investigators will follow the participant during and after the injections. To learn more about the way the T cells are working in the participant's body, up to 60 mL (upto 12 teaspoons, no more than 3ml/kg/day) of blood will be taken from the participant before the chemotherapy, before the T-cell infusion, 1 to 4 hours after the infusion, 3 to 4 days after the infusion (this time point is optional ) at 1 week, 2 weeks, 4 weeks and 8 weeks after the injection, every 3 months for 1 year, every 6 months for 4 years and then every year for the next 10 years. Total participation time for this study will be 15 years.

During the time points listed above, if the T cells are found in the participant's blood at a certain amount an extra 5 mL of blood may need to be collected for additional testing.

The investigators will use this blood to look for the frequency and activity of the cells that the investigators have given; that is, to learn more about the way the T cells are working and how long they last in the body. The investigators will also use this blood to see if there are any long-term side effects of putting the new gene (chimeric antigen receptor, CAR) into the cells. In addition to the blood draws, because the participants have received cells that have had a new gene put in them, the participants will need to have long term follow up for 15 years so the investigators can see if there are any long-term side effects of the gene transfer.

Once a year, the participants will be asked to have their blood drawn and answer questions about their general health and medical condition. The investigators may ask the participants to report any recent hospitalizations, new medications, or the development of conditions or illness that were not present when the participants enrolled in the study and may request that physical exams and/or laboratory tests be performed if necessary.

When tumor biopsy is performed for clinical reasons the investigators will request permission to obtain excess sample to learn more about the effects of the treatment on the participant's disease.

In the event of death, the investigators will request permission to perform an autopsy to learn more about the effects of the treatment on the participant's disease and if there were any side effects from the cells with the new gene.

In addition, the investigators would like to ask for participant permission to use tumor biopsy for research purposes only. Associated risk with the biopsy will be discussed with each participant in detail in a procedure specific consent form. The investigators will test the sample to see if the GAP T cells can be found in the tumor and what effect they had on the tumor cells.

If participants develop a second abnormal cancer growth, significant blood or nervous system disorder during the trial, a biopsy sample of the tissue will be tested.

ELIGIBILITY:
Procurement Eligibility

Inclusion Criteria:

* Relapsed or refractory GPC3-positive* solid tumors (currently only enrolling liver tumors)
* Age ≥ 1 year and ≤ 21 years
* Lansky or Karnofsky score ≥60%
* Life expectancy ≥16 weeks
* Child-Pugh-Turcotte score <7 (for patients with hepatocellular carcinoma only)
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

Exclusion Criteria:

* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies)
* History of organ transplantation
* Known HIV positivity
* Active bacterial, fungal or viral infection (except Hepatitis B or Hepatitis C virus infections)
* Severe previous toxicity from cyclophosphamide or fludarabine

Treatment Eligibility

Inclusion Criteria:

* Age ≥ 1 year and ≤ 21 years
* Barcelona Clinic Liver Cancer Stage A, B or C (for patients with hepatocellular carcinoma only)
* Life expectancy of ≥ 12 weeks
* Lansky or Karnofsky score ≥ 60%
* Child-Pugh-Turcotte score < 7 (for patients with hepatocellular carcinoma only)
* Adequate organ function:

  * Creatinine clearance as estimated by Cockcroft Gault or Schwartz ≥ 60 ml/min
  * serum AST< 5 times ULN
  * total bilirubin < 3 times ULN for age
  * INR ≤1.7 (for patients with hepatocellular carcinoma only)
  * absolute neutrophil count > 500/microliter
  * platelet count > 25,000/microliter (can be transfused)
  * Hgb ≥7.0 g/dl (can be transfused)
  * pulse oximetry >90% on room air
* Recovered from acute toxic effects of all prior chemotherapy and investigational agents before entering this study
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 3 months after the T-cell infusion.
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

Exclusion Criteria

* Pregnancy or lactation
* Uncontrolled infection
* Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day, dose adjustment or discontinuation of medication must occur at least 24 hours prior to CAR T cell infusion)
* Known HIV positivity
* Active bacterial, fungal or viral infection (except Hepatitis B or Hepatitis C virus infections)
* History of organ transplantation
* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies)
* Severe previous toxicity from cyclophosphamide or fludarabine

GPC3 expression will be evaluated by standard immunohistochemistry (IHC). A tumor is considered GPC3 positive, when the staining is Grade 2 (>25% positive tumor cells) or above with an intensity score of 2 or above on a scale of 0 to 4.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2037-02 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | 6 weeks
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the GPC3-CAR T cells. Specifically those which are Grade 5; non-hematologic Grade 3-4 not returning to Grade 2 within 72 hours; Grade 2-4 allergic reaction; Hematologic Grade 4 that fails to return to Grade 2 or baseline (whichever is more severe) within 14 days; all grade 4 CRS and neurologic toxicities and grade 3 CRS and neurologic toxicities that fail to return to Grade 1 within 7 days.

SECONDARY OUTCOMES:
Percent of Patients with best response as either complete remission or partial remission | 6 weeks
  Response rates will be estimated as the percent of patients whose best response is either complete remission or partial remission by combining the data from the two patients. To compare with historical data, a 95% confidence interval will be calculated for the response rate.
Median T cell persistence | 15 years
  as measured by PCR

CONTACTS AND LOCATIONS:
Overall Officials: David Steffin, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No